CLINICAL TRIAL: NCT01187953
Title: Ph3,DB/DD,Multi-Ctr,Pros,Rand Study-Efficacy and Safety of LCP-Tacro™ Tablets, QD, Compared to Prograf® Capsules,BID, in Combination With Mycophenolate Mofetil for Acute Allograft Rejection in De Novo Kidney Transplant
Brief Title: Double-Blind,Double-Dummy,Efficacy/Safety,LCP-Tacro™ Vs Prograf®,Prevention Rejection,De Novo Adult Kidney Tx
Acronym: LCPTacro3002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LCP-Tacro-3002
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Renal Failure
Keywords: Tacrolimus; Acute Rejection; Kidney
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCP-Tacro (Experimental): The initial dose of 0.17 mg/kg will be administered orally in the morning (before noon) within 24 hours following transplantation. Subsequent doses will be adjusted according to whole blood tacrolimus trough levels.
  Interventions: Drug: LCP-Tacro
- Prograf (tacrolimus) (Experimental): Starting total daily dose of 0.10 mg/kg administered in two equally divided doses, morning and evening, per product labeling. Doses will be adjusted according to whole blood tacrolimus trough levels. In the initial post-transplant period, plasma trough levels will be measured at 24 and 48 hours. Study drugs will be adjusted to maintain the whole blood pre-dose (trough) concentration of tacrolimus in the target range of 6 - 11 ng/mL for the first 30 days, then 4 - 11 ng/mL for the remainder of the study.
  Interventions: Drug: Prograf (tacrolimus)

INTERVENTIONS:
Drug: Prograf (tacrolimus) — Administered per current product labeling
  Other Names: tacrolimus
  Arms: Prograf (tacrolimus)
Drug: LCP-Tacro — Tacrolimus, once-per-day The initial dose of 0.17 mg/kg will be administered orally in the morning (before noon) within 24 hours following transplantation. Subsequent doses will be adjusted according to whole blood tacrolimus trough levels.
  Other Names: Tacrolimus modifed-release
  Arms: LCP-Tacro

SUMMARY:
This study will evaluate the efficacy and safety of LCP-Tacro (tacrolimus) Tablets administered once-a-day compared to Prograf (tacrolimus) Capsules twice-a-day as immunosuppression for the prevention of organ rejection in newly transplanted adult kidney transplant recipients. Patients will be treated for a 12 month study period followed by a 12 month, blinded extension treatment period To show that LCP-Tacro Tablets are clinically similar to Prograf Capsules in the prevention of acute rejection.

DETAILED DESCRIPTION:
This is a two-armed parallel group, prospective, randomized, double-blind, double-dummy,multicenter Phase 3 clinical study to establish the efficacy and safety of LCP-Tacro Tablets (tacrolimus, LifeCycle Pharma A/S, Hørsholm, Denmark) once daily for the prevention of allograft rejection in de novo adult male and female recipients of a primary or secondary kidney transplant evaluated by a combined efficacy endpoint comprised of acute rejection, graft loss and patient loss. The trial is designed to determine if the test drug, LCP-Tacro, is not inferior to an unacceptable extent to the reference compound, Prograf. Recipients of a kidney transplant who sign an informed consent form and fulfill all other inclusion and exclusion criteria will be randomly assigned to once-daily therapy with LCP-Tacro Tablets or to twice-daily therapy with Prograf Capsules (tacrolimus, Astellas Pharma US, Inc., Deerfield, IL), each concomitantly administered with mycophenolate mofetil (MMF) and corticosteroids. All patients will also receive interleukin-2 (IL-2) receptor antagonist (e.g.,Simulect®, basiliximab; Novartis Pharmaceuticals, East Hanover, NJ). Following screening,transplantation, and randomization, study visits will be conducted over a 12-month treatment period; with additional visits during a 12 month extension period on treatment and a follow-up safety assessment by visit or telephone interview 30 days after withdrawal from study drug.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. 18 and 70 years, inclusive
3. receiving primary or secondary renal allograft from a deceased donor or non-human leukocyte antigen (HLA) identical living donor
4. no known contraindications to the administration of IL-2 receptor antagonist induction therapy, MMF, corticosteroids or tacrolimus
5. negative pregnancy test
6. Negative cross match test, and compatible (A, B, AB or O) blood type
7. Able to swallow tablets and capsules

Exclusion Criteria:

1. Recipients of any non-renal transplant (solid organ or bone marrow) ever
2. Panel reactive antibody (PRA) >30%
3. Patients with any condition that may affect study drug absorption (e.g. gastrectomy or clinically significant diabetic gastroenteropathy)
4. Body mass index (BMI) 18 kg/m2
5. History of alcohol abuse
6. History of recreational drug abuse
7. Screening 12-lead electrocardiogram (ECG) demonstrating clinically relevant abnormalities
8. WOCBP who are either pregnant, lactating, planning to become pregnant
9. Patients with an oral temperature (prior to study drug dosing) of 38.0 ºC (100.4 ºF) or higher
10. Patients with clinically significant active infections
11. Patients with a known hereditary immunodeficiency
12. Patients with malignancies or with a history of malignancies (within the last 5 years)
13. Patients who are receiving or expect to receive sirolimus, everolimus, azathioprine,or cyclophosphamide within 3 months prior to enrollment
14. Patients with evidence of clinically significant disease (e.g., cardiac, gastrointestinal or hepatic disorders)
15. Patients with reversible cardiac ischemia (history of untreated reversible ischemia on stress test)
16. Patients with clinically symptomatic congestive heart failure or documented ejection fraction of less than 45%
17. Patients with significant chronic obstructive pulmonary disease, pulmonary restrictive disease or significant pulmonary hypertension
18. Treatment with an investigational drug, device or regimen within 1 year preceding the first dose of study drug
19. Patients who are unwilling to refrain from consumption of grapefruit or grapefruit containing juices
20. Patients receiving concomitant drugs that may affect concentrations of tacrolimus in whole blood, as listed in Appendix 2
21. Laboratory variables that are abnormal (outside laboratory reference range) and clinically relevant, as judged by the Investigator
22. Patients with positive results of any of the following serological tests: human immunodeficiency virus (HIV)-1 antibody, hepatitis B virus (HBV) surface antigen (HBsAg), anti-hepatitis B core antibody (HBcAb), and anti-hepatitis C virus (HCV)antibody (HCV Ab).
23. Patients who experienced graft loss within 1 year of transplant, due to acute rejection or due to BK nephropathy
24. Patients having experienced focal segmental glomerulosclerosis (FSGS)
25. Donor with positive serological test result for HIV-1, HBV or HCV
26. Donor with history of malignant disease (current or historical)
27. Centers for Disease Control and Prevention high-risk donor
28. Patients with mental dysfunction or inability to cooperate with the study
29. Cold ischemia time >30 hours

29. Non-heart-beating donor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Glicklich, Study Director — VP, Clinical Operations
Locations (86):
- United States (46):
  - Clinical Site 1020, Birmingham, Alabama
  - Clinical Site 1031, Loma Linda, California
  - Clinical Site 1009, Los Angeles, California
  - Clinical Site 1022, Sacremento, California
  - Clinical Site 1045, San Diego, California
  - Clinical Site 1049, San Diego, California
  - Clinical Site 1044, San Francisco, California
  - Clinical Site 1011, Denver, Colorado
  - Clinical Site 1003, New Haven, Connecticut
  - Clinical Site 1036, Gainesville, Florida
  - Clinical Site 1013, Miami, Florida
  - Clinical Site 1038, Orlando, Florida
  - Clinical Site 1006, Tampa, Florida
  - Clinical Site 1055, Atlanta, Georgia
  - Clinical Site 1053, Chicago, Illinois
  - Clinical Site 1056, Peoria, Illinois
  - Clinical Site 1026, New Orleans, Louisiana
  - Clinical Site 1052, Portland, Maine
  - Clinical Site 1014, Boston, Massachusetts
  - Clinical Site 1018, Detroit, Michigan
  - Clinical Site 1048, Hackensack, New Jersey
  - Clinical Site 1037, Livingston, New Jersey
  - Clinical Site 1033, New Brunswick, New Jersey
  - Clinical Site 1060, Albany, New York
  - Clinical Site 1042, Buffalo, New York
  - Clinical Site 1040, East Setauket, New York
  - Clinical Site 1050, New York, New York
  - Clinical Site 1019, New York, New York
  - Clinical Site 1025, New York, New York
  - Clinical Site 1035, The Bronx, New York
  - Clinical Site 1010, Valhalla, New York
  - Clinical Site 1051, Chapel Hill, North Carolina
  - Clinical Site 1032, Durham, North Carolina
  - Clinical Site 1058, Greenville, North Carolina
  - Clinical Site 1005, Cleveland, Ohio
  - Clinical Site 1054, Harrisburg, Pennsylvania
  - Clinical Site 1023, Philadelphia, Pennsylvania
  - Clinical Site 1021, Providence, Rhode Island
  - Clinical Site 1012, Charleston, South Carolina
  - Clinical Site 1047, Nashville, Tennessee
  - Clinical Site 1029, Houston, Texas
  - Clinical Site 1061, San Antonio, Texas
  - Clinical Site 1039, San Antonio, Texas
  - Clinical Site 1027, Richmond, Virginia
  - Clinical Site 1046, Madison, Wisconsin
  - Clinical Site 1008, Milwaukee, Wisconsin
- Argentina (2):
  - Clinical Site 54163, Buenos Aires
  - Clinical Site 54164, Córdoba
- Australia (6):
  - Clinical Site 61101, Camperdown, New South Wales
  - Clinical Site 61105, Woodville, South Australia
  - Clinical Site 61100, Clayton, Victoria
  - Clinical Site 61104, Parkville, Victoria
  - Clinical Site 61102, Nedlands, Western Australia
  - Clinical Site 61106, Perth, Western Australia
- Brazil (6):
  - Clinical Site 55178, Juiz de Fora
  - Clinical Site 55172, Porto Alegre, Rio Grande Do Sul
  - Clinical Site 55179, Porto Alegre, Rio Grande Do Sul
  - Clinical Site 55175, Ribeirão Preto
  - Clinical Site 55173, Rio de Janeiro
  - Clinical Site 55171, São Paulo
- France (4):
  - Clinical Site 33132, Brest
  - Clinical Site 33131, Nice
  - Clinical Site 33136, Saint-Etienne
  - Clinical Site 33134, Toulouse
- Germany (2):
  - Clinical Site 49137, Berlin
  - Clinical Site 49139, Essen
- Clinical Site 39144, Roma, Italy
- Mexico (4):
  - Clinical Site 52184, Aguascalientes
  - Clinical Site 52181, Cuernavaca, MOR
  - Clinical Site 52183, Mexico City
  - Clinical Site 52182, Mexico City
- New Zealand (2):
  - Clinical Site 64112, Auckland
  - Clinical Site 64121, Wellington South
- Poland (3):
  - Clinical Site 48151, Bydgoszcz
  - Clinical Site 48148, Szczecin
  - Clinical Site 48149, Warsaw
- Serbia (3):
  - Clinical Site 381140, Belgrade
  - Clinical Site 381141, Niš
  - Clinical Site 381142, Novi Sad
- Singapore (2):
  - Clinical Site 65127, Singapore
  - Clinical Site 65126, Singapore
- Clinical Site 92113, Seoul, South Korea
- Spain (3):
  - Clinical Site 34155, Barcelona, Catalonia
  - Clinical Site 34157, Barcelona, Catalonia
  - Clinical Site 34151, L'Hospitalet de Llobregat, Catalonia
- Clinical Site 46161, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Started | 268 | 275
Dosed | 266 | 271
Completed | 253 | 254
Not Completed | 15 | 21
Not completed — Death | 11 | 13
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: The patient sample was predominantly White (76.8%) and male (65.4%).
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-Tacro | Prograf (Tacrolimus) | Total
Number analyzed (Participants) | 268 | 275 | 543
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 247 | 499
  >=65 years | 16 | 28 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.29) | 46.9 (14.26) | 45.8 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 94 | 188
  Male | 174 | 181 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 79 | 153
  Not Hispanic or Latino | 194 | 196 | 390
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 15 | 25
  White | 203 | 214 | 417
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 44 | 34 | 78
Region of Enrollment [Number; unit: participants]
  Argentina | 1 | 1 | 2
  Singapore | 1 | 1 | 2
  United States | 67 | 70 | 137
  Spain | 24 | 21 | 45
  New Zealand | 2 | 3 | 5
  Poland | 27 | 26 | 53
  Brazil | 29 | 29 | 58
  Mexico | 27 | 29 | 56
  Italy | 6 | 6 | 12
  Australia | 11 | 11 | 22
  France | 35 | 38 | 73
  Serbia | 6 | 5 | 11
  Germany | 32 | 35 | 67
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.72 (4.648) | 26.68 (4.948) | 26.21 (4.822)
Diabetes at the time of transplant [Number; unit: participants]
  Patients with diabetes at transplant | 50 | 56 | 106
  Patients without diabetes at transplant | 218 | 219 | 437
Time from transplant to first dose [Mean (Standard Deviation); unit: hours] | 34.15 (8.878) | 34.38 (9.735) | 34.27 (9.312)
Donor Type [Number; unit: participants]
  Living | 135 | 129 | 264
  Deceased | 133 | 145 | 278
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint for the Study is the Proportion of Treatment Failures Within 12 Months After Randomization to Study Drug.
Description: Treatment failure is a composite endpoint; a patient is considered a treatment failure if the patient experienced any of the following events during this period: death, graft failure, BPAR (Banff grade ≥1A) or lost to follow-up.
Time Frame: 360 days
Population: All 543 randomized patients were included in the analysis population.
Measure: Number; unit: participants
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 268 | 275
participants
  Death | 8 | 8
  Graft Failure | 9 | 11
  Biobsy Proven Acute Rejection | 35 | 37
  Lost to follow up | 4 | 5
Statistical Analysis 1: Comparison: LCP-Tacro vs Prograf (Tacrolimus); No overall p value was calculated, only individual p values for each endpoint category. One statistical analysis table is reported for each individual p value; Test type: Non-Inferiority or Equivalence — It was assumed that both treatment groups in this study would have a 15% 12-month treatment failure rate, the study will require 270 patients per group to have 90% power to reject the null hypothesis that the investigational drug, LCP-tacro, is inferior to the reference drug, Prograf, based on a 2-sided 95% CI for the difference and a 0.10 non-inferiority margin; p > 0.999, Fisher Exact — Endpoint: Death
Statistical Analysis 2: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.821, Fisher Exact — Endpoint: Graft Failure
Statistical Analysis 3: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.900, Fisher Exact — Endpoint: BPAR
Statistical Analysis 4: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.999, Fisher Exact — Endpoint: Lost to follow up

2. Secondary Outcome: For the 24-month Analysis, the Endpoint Includes Additional Treatment Failures That Occurred During the 12-month Treatment Extension Period, up to Day 734 After the Randomization Date.
Description: Treatment failure is a composite endpoint; a patient is considered a treatment failure if the patient experienced any of the following events during this period (day 1 to day 734): death, graft failure, BPAR (Banff grade ≥1A) or lost to follow-up.
Time Frame: 734 days
Population: All 543 randomized patients were included in the analysis population.
Measure: Number; unit: participants
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 268 | 275
participants
  Death | 11 | 13
  Graft Failure | 11 | 15
  Biobsy Proven Acute Rejection | 46 | 50
  Lost to follow up | 4 | 8
Statistical Analysis 1: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.835, Fisher Exact — Endpoint: Death
Statistical Analysis 2: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.548, Fisher Exact — Endpoint: Graft Failure
Statistical Analysis 3: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.822, Fisher Exact — Endpoint: BPAR
Statistical Analysis 4: Comparison: LCP-Tacro vs Prograf (Tacrolimus); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.383, Fisher Exact — Endpoint: Lost to follow up

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day of first dose of study drug and up until 30 days after completing the 24 months study period.
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Serious Adverse Events (participants affected / at risk) | 166/268 | 185/275
Other Adverse Events (participants affected / at risk) | 263/268 | 269/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=268) | Prograf (Tacrolimus) (N=275)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemolytic Anaemie (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 1 (2) | 3 (3)
Cardiac Failure (Cardiac disorders) | 2 (3) | 2 (5)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (2)
Coronary artery stenosis (Cardiac disorders) | 9 (9) | 1 (1)
Tachyarrhytmia (Cardiac disorders) | 0 (0) | 1 (1)
Aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gatritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (3)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroinstestinal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2) | 0 (0)
Intestinal Ischaemie (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 1 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site erosion (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Organ Failure (General disorders) | 1 (1) | 0 (0)
Cholesystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 23 (28) | 33 (39)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Pancreas transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 26 (34) | 22 (41)
Cytomegalovirus infection (Infections and infestations) | 12 (13) | 10 (12)
Pneumonia (Infections and infestations) | 4 (5) | 10 (10)
Gastroenteritis (Infections and infestations) | 9 (10) | 3 (3)
Pyelonephritis (Infections and infestations) | 7 (8) | 5 (6)
Sepsis (Infections and infestations) | 5 (8) | 6 (10)
Urosepsis (Infections and infestations) | 6 (7) | 5 (6)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 2 (4) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 2 (2)
Polyomavirus-associated nephropathy (Infections and infestations) | 3 (5) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 2 (3)
Herpes Zoster (Infections and infestations) | 1 (1) | 1 (1)
Herpes Zoster disseminated (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Adenoviral haemorrhagic cystitis (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitits (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitits bacterial (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Human polyomavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (2)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Prostatitis escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Urinary baldder abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Wound Abscess (Infections and infestations) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 8 (8) | 18 (18)
Graft dysfunction (Injury, poisoning and procedural complications) | 7 (12) | 7 (9)
Transplant failure (Injury, poisoning and procedural complications) | 4 (6) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 2 (5)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Graft Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Graft Complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Shunt Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle frature (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve replacement complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perirenal kaematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post precedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 8 (9) | 13 (17)
Liver function test abnormal (Investigations) | 0 (0) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Immunosuppressant drug level increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadeqaute control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extrenities (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Aubarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 1 (1) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (3)
Suicidal attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 12 (19)
Renal impairment (Renal and urinary disorders) | 4 (4) | 6 (7)
Renal artery stenosis (Renal and urinary disorders) | 3 (3) | 3 (4)
Ureteric artery stenosis (Renal and urinary disorders) | 3 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 4 (4) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (5) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal artery Thrombosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Ureteral necrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 2 (3)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 1 (4) | 1 (1)
Renal cyst ruptures (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal vein thrombosis (Renal and urinary disorders) | 1 (2) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (2) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (3) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (2) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolaps (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pregnancy partner (Social circumstances) | 0 (0) | 1 (1)
Lymphocele marsipialisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 3 (4) | 9 (15)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 3 (7) | 0 (0)
Arterial thrombosis (Vascular disorders) | 2 (7) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Extrinsic iliac vein compression (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=268) | Prograf (Tacrolimus) (N=275)
Anaemia (Blood and lymphatic system disorders) | 75 (91) | 84 (98)
Leukopenia (Blood and lymphatic system disorders) | 37 (43) | 39 (42)
Polycythaemia (Blood and lymphatic system disorders) | 17 (22) | 19 (22)
Diarrhoea (Gastrointestinal disorders) | 91 (125) | 102 (159)
Constipation (Gastrointestinal disorders) | 51 (56) | 68 (81)
Nausea (Gastrointestinal disorders) | 40 (57) | 43 (52)
Abdominal pain (Gastrointestinal disorders) | 24 (28) | 33 (40)
Vomiting (Gastrointestinal disorders) | 17 (22) | 26 (30)
Dyspepsia (Gastrointestinal disorders) | 19 (20) | 19 (21)
Abdominal pain upper (Gastrointestinal disorders) | 14 (18) | 14 (15)
Oedema peripheral (General disorders) | 50 (78) | 66 (90)
Pyrexia (General disorders) | 23 (27) | 21 (25)
Asthenia (General disorders) | 14 (15) | 13 (15)
Kidney transplant rejection (Immune system disorders) | 38 (49) | 45 (55)
Urinary tract infection (Infections and infestations) | 81 (136) | 80 (169)
BK virus infection (Infections and infestations) | 23 (28) | 29 (34)
Upper respiratory tract infection (Infections and infestations) | 30 (39) | 21 (26)
Nasopharyngitis (Infections and infestations) | 26 (30) | 18 (21)
Cytomegalovirus infection (Infections and infestations) | 21 (26) | 18 (27)
Gastroenteritis (Infections and infestations) | 21 (25) | 13 (14)
Sinusitis (Infections and infestations) | 13 (17) | 19 (25)
Bronchitits (Infections and infestations) | 18 (18) | 12 (16)
Complications of kidney transplant (Injury, poisoning and procedural complications) | 20 (23) | 30 (33)
Wound complication (Injury, poisoning and procedural complications) | 20 (24) | 18 (21)
Procedural pain (Injury, poisoning and procedural complications) | 14 (15) | 19 (21)
Blood creatinine increased (Investigations) | 33 (44) | 39 (53)
Weight increased (Investigations) | 21 (25) | 22 (23)
Diabetes mellitus (Metabolism and nutrition disorders) | 55 (64) | 42 (49)
Hypophosphataemia (Metabolism and nutrition disorders) | 36 (45) | 42 (46)
Hyperkalaemia (Metabolism and nutrition disorders) | 42 (52) | 34 (40)
Hypokalaemia (Metabolism and nutrition disorders) | 34 (38) | 37 (46)
Hyperglycemia (Metabolism and nutrition disorders) | 31 (34) | 37 (42)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (41) | 33 (39)
Vitamin D deficiency (Metabolism and nutrition disorders) | 27 (28) | 27 (29)
Hypucalcaemia (Metabolism and nutrition disorders) | 21 (23) | 25 (25)
Dyslipidaemia (Metabolism and nutrition disorders) | 23 (24) | 17 (19)
Metabolic acidosis (Metabolism and nutrition disorders) | 22 (24) | 16 (18)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 (17) | 16 (16)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (10) | 20 (21)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (17) | 16 (16)
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 (14) | 15 (15)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14 (15) | 15 (16)
Dehydration (Metabolism and nutrition disorders) | 14 (17) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (24) | 18 (22)
Pain in extrimity (Musculoskeletal and connective tissue disorders) | 22 (25) | 17 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 14 (17)
Tremor (Nervous system disorders) | 59 (66) | 51 (60)
Headache (Nervous system disorders) | 43 (54) | 29 (41)
Dizziness (Nervous system disorders) | 19 (21) | 14 (18)
Insomnia (Psychiatric disorders) | 38 (42) | 29 (32)
Anxiety (Nervous system disorders) | 24 (28) | 25 (30)
Renal impairment (Renal and urinary disorders) | 20 (23) | 27 (37)
Proteinuria (Renal and urinary disorders) | 19 (20) | 21 (24)
Haematuria (Renal and urinary disorders) | 18 (20) | 20 (23)
Dysuria (Renal and urinary disorders) | 20 (26) | 15 (15)
Renal failure acute (Renal and urinary disorders) | 12 (13) | 17 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (29) | 30 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 21 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (19) | 21 (23)
Acne (Skin and subcutaneous tissue disorders) | 17 (18) | 19 (20)
Hypertension (Vascular disorders) | 71 (81) | 73 (88)
Hypotension (Vascular disorders) | 20 (21) | 15 (18)
Lymphocele (Vascular disorders) | 5 (6) | 15 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other